CLINICAL TRIAL: NCT03503396
Title: Risk for Alcohol Impaired Driving: From the Laboratory to the Natural Environment
Brief Title: Alcohol Impaired Driving in the Natural Environment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Denis McCarthy, Professor, University of Missouri-Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2010187; R01AA019546-06A1 (NIH)
Record Dates: First submitted 2018-04-11; First posted 2018-04-19 (Actual); Results first posted 2023-05-03 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-04

CONDITIONS: Driving Under the Influence
Keywords: drunk driving; alcohol impaired driving; drinking and driving; ambulatory assessment
MeSH Terms: conditions — Driving Under the Influence

STUDY DESIGN:
Intervention Model Description: Participants will be assigned to either receive feedback from a breathalyzer device or to receive no information.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BAC feedback (Experimental): Participants will receive a warning when their BAC is above a set limit (cutpoint is not disclosed by well below legal limit). Warning will notify them that their results indicate it is not safe for them to drive.
  Interventions: Behavioral: BAC Driving Feedback/Warning
- No Feedback (Active Comparator): Participants will not receive any information on their BAC from their device.
  Interventions: Behavioral: No Feedback

INTERVENTIONS:
Behavioral: BAC Driving Feedback/Warning — Participants will receive a warning at a set BAC limit, indicating they are too impaired to drive.
  Arms: BAC feedback
Behavioral: No Feedback — Participants will receive no information about BAC, but will still complete study assessments and provide breath samples during drinking sessions.
  Arms: No Feedback

SUMMARY:
This is a pilot study to set up a larger investigation examining predictors of the decision to drive after consuming alcohol. All participants will carry a study provided smartphone and breathalyzer device for the 2 week period of the study. The intervention is that participants are randomly assigned to one of 2 breathalyzer feedback conditions - one where they receive a warning that their results indicate they should not drive and one where they receive no feedback. The study is designed to provide information needed for a larger version with a similar protocol, but also to provide an initial test of project hypotheses as well.

DETAILED DESCRIPTION:
Despite previous success in reducing alcohol impaired driving (AID) and fatal crashes, rates have not decreased significantly since the 1990s. Developing novel approaches to prevention/intervention are likely required to produce further progress.

This project is designed to evaluate a potential intervention for AID using mobile technology. In addition, the project is designed to provide pilot data for a large scale investigation.

Recent laboratory work by the PI has demonstrated the utility of assessing AID risk factors when participants are intoxicated. We identified four risk factors that, measured under intoxication, are cross-sectional predictors of AID: AID attitudes (Morris et al., 2014), impulsivity (McCarthy et al., 2012), behavioral economic demand (Amlung et al., 2016) and subjective intoxication (Amlung et al., 2014).

The proposed project will evaluate these factors as prospective predictors of AID and extend this work outside the laboratory and into participants' natural drinking environment using Ambulatory Assessment (AA). AA is a set of techniques used to collect data from individuals in the course of their daily life. AA methods provide increased ecological validity across multiple modalities (e.g., self-report, physiological measures). No study to date has used AA to examine AID. We will employ a combination of three AA methods: ecological momentary assessment, geospatial technology, and portable breath analysis.

Ecological Momentary Assessment (EMA) is a form of AA that allows participants to self-report on their current thoughts, feelings, and behaviors in their natural environment (Shiffman et al., 2008). EMA avoids most pitfalls of retrospective reports, and is increasingly used to study temporally proximal influences on substance use behaviors (Shiffman, 2009). Despite the importance of such influences to AID decisions (Quinn & Fromme, 2012), no study to date has applied EMA methods to the study of AID.

Advancements in mobile technology, such as global position systems (GPS) and portable breathalizers, allow for the collection of objective data on participant location and alcohol use in real-time. We will combine location data (e.g., drinking venue, distance from home) and in-the-moment breathalyzer data with self-report EMA data from each participant drinking episode. This combination will allow for a more complete assessment of event-level factors that contribute to AID decisions.

This pilot project will test the hypothesis that temporally proximal measures of AID risk factors (subjective impairment, perceived risk) collected during a drinking episode will improve prediction of AID, over and above trait measures of AID risk factors.

The pilot project will also test the potential for AA to function as an intervention for AID. In this pilot, participants will be randomly assigned to either receive some feedback from their breathalyzer (a warning that they have consumed too much to drive safely) or not to receive any feedback. Note that participants will not be told their BAC, due to potential risks of specific feedback (increased consumption, titrating drinking to drive at slightly below .08). Instead, feedback will be general ("Your results indicate that you have drank too much to drive safely"), and participants will not be aware of what BAC triggers these warnings.

Comparisons of all participants AID behavior at baseline (from a Timeline Follow-back assessment) with their AID behavior during study participation will be used to test whether the increased self-monitoring of AA can alter AID decisions. In addition, comparisons between groups (feedback vs. none) will test for potential effects of BAC feedback on AID decisions. Support for these hypotheses could lead to novel, cost-effective interventions to reduce AID using mobile technology.

This pilot will enroll 40 moderate-to-heavy drinking young adults. Participants will complete a brief laboratory session of AID risk measures, followed by two weeks of AA. They will be randomly assigned to one of two conditions (BAC feedback vs. none). Interview assessments of AID will be conducted at baseline and at the completion of AA assessments, with interviewers blind to condition.

ELIGIBILITY:
Inclusion Criteria:

* moderate to heavy drinkers.
* must drive regularly (including driving for social events).
* report binge drinking (4/5 drinks in a 2 hour period) at least once in the past month
* fluent in english

Exclusion Criteria:

* no exclusion criteria other than failure to meet inclusion criteria

Ages: 21 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2018-04-02 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-01-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Missouri-Columbia, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | BAC Feedback | No Feedback
Started | 24 | 24
Completed | 22 | 24
Not Completed | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BAC Feedback | No Feedback | Total
Number analyzed (Participants) | 24 | 24 | 48
Age, Continuous [Mean (Full Range); unit: years] | 22.75 [21 to 28] | 22.66 [21 to 27] | 22.71 [21 to 28]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 19 | 35
  Male | 8 | 5 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 24 | 24 | 48
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 4 | 6
  White | 21 | 17 | 38
  More than one race | 1 | 3 | 4
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 24 | 24 | 48

OUTCOME MEASURES:

1. Primary Outcome: Alcohol Impaired Driving Behavior
Description: Change in number of times driven after drinking per week from pre (4 week TLFB) to post (2 week TLFB). A Timeline Followback (TLFB) is an interview where the participant self-reports their drinking behavior including: where they were drinking, how much they drank of what over what period of time, what location they went to next, how they got there.
Time Frame: Baseline (4 week prior to initial interview) and trial period (2 weeks after initial interview)
Measure: Number; unit: Count of driving episodes after drinking
Arm/Group | BAC Feedback | No Feedback
Number analyzed (Participants) | 24 | 24
Count of driving episodes after drinking
  Baseline | 67 | 60
  Trial period | 36 | 29

2. Secondary Outcome: Perceived Risk of Driving After Drinking
Description: Rating of danger of driving after receiving warning. Participants were asked to rate the perceived dangerousness of driving during drinking episodes by asking them to "indicate how dangerous you feel it would be for you to drive "right now"" Responses are recorded on a 1 (not at all dangerous) to 10 (extremely dangerous) visual analogue scale.
Time Frame: Self-reported current perception (i.e., "right now")
Measure: Mean (95% Confidence Interval); unit: score on a scale (1-10)
Arm/Group | BAC Feedback | No Feedback
Number analyzed (Participants) | 23 | 22
score on a scale (1-10) | 2.9176 [1.6895 to 4.1456] | 1.6705 [0.9651 to 2.3758]

3. Other Pre Specified Outcome: Proximal Predictors of Impaired Driving
Description: Outside of the intervention effect, observational data will be used to test hypotheses about proximal predictors of driving behavior.
Time Frame: 2 weeks of study intervention
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Effect of Self-monitoring on AID Behavior and Perceptions
Description: Outside of the intervention effect, observational data will be used to test hypotheses about whether all participants report reduced driving after drinking and increase perceive risk of driving after drinking during the intervention period.
Time Frame: 2 weeks of study intervention
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Two weeks
Arm/Group | BAC Feedback | No Feedback
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 0/24 | 0/24

LIMITATIONS AND CAVEATS:
Due to the relatively brief EMA data collection period in this pilot/feasibility study, few alcohol-impaired driving events occurred during the study period, and we instead focused on driving intentions as the primary outcome.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-12-03): https://cdn.clinicaltrials.gov/large-docs/96/NCT03503396/Prot_SAP_000.pdf
  • Informed Consent Form (2018-02-27): https://cdn.clinicaltrials.gov/large-docs/96/NCT03503396/ICF_001.pdf